CLINICAL TRIAL: NCT06196164
Title: A Randomized Controlled Trial of Malignancy Low Biliary Tract Obstruction Drainage Strategies
Brief Title: A RCT of Low MBO Drainage Strategies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wu Xi, associate professor，M.D., Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K3807
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Jaundice, Obstructive; Cholangiopancreatography, Endoscopic Retrograde; Endoscopic Ultrasound-Guided Drainage
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-BD (Experimental): Endoscopic Ultrasound-guided Biliary Drainage
  Interventions: Procedure: EUS-BD
- ERCP-BD (Other): Endoscopic Retrograde Cholangiopancreatography
  Interventions: Procedure: ERCP-BD

INTERVENTIONS:
Procedure: EUS-BD — We observe the bile duct through endoscopic ultrasound, then puncture through the gastric or duodenum wall and place a guide wire, expanding along the guide wire, finally place a stent between the bile duct and the stomach or intestine for drainage.
  Arms: EUS-BD
Procedure: ERCP-BD — We use a Duodenoscopy to pass through mouth down to the small opening where the bile duct and pancreatic drain. A small narrow catheter is passed through the scope to gain access to the drainage duct , followed by advancement of a wire deep into the duct. A small cut is made at the bile duct opening to help facilitate a stent placed in the bile duct.
  Arms: ERCP-BD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of EUS-BD compared with ERCP-BD in low biliary obstruction caused by periampullary cancer, pancreatic cancer or low bile duct cancer. This is a single center, prospective, randomized-controlled study. The primary endpoint of this study is stent patency time, and secondary endpoints include technical success rate, clinical success rate, operation time, operation related complications rate, reintervention rate, stent patency rate at 6 months, and 1-year postoperative survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 years old or above;
2. Periampullary cancer/pancreatic cancer according to pathology or clinical judgment of more than 2 senior doctors;
3. Distal malignant bile duct obstruction (2cm away from the hepatic hilum);
4. Ultrasound evaluation shows that the accessible part of the bile duct has a width of ≥ 12mm;
5. The patient or family member is able to understand the research protocol and is willing to participate in this study, providing written informed consent.

Exclusion Criteria:

1. Patients suffer from severe cardiovascular or pulmonary diseases who are unable to tolerate anesthesia or endoscopic examination;
2. Uncorrectable coagulation abnormalities or bleeding tendencies (INR>1.5 or platelets<50) × 109 /L);
3. There is a plan for subsequent surgical resection of the tumor, accompanied by severe infection or an expected survival period of less than 3 months;
4. Successful biliary drainage measures have been implemented, including but not limited to ERCP, ENBD, PTCD, and surgical procedures;
5. Previous surgical changes to the anatomical structure of the pancreas, gallbladder, stomach, and duodenum;
6. Pregnancy, lactation, or planned pregnancy;
7. Refusal to join or inability to provide informed consent;
8. Other researchers evaluated the unsuitability of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
stent patency time | 0-24months
  The interval between the operation day and the occurrence of cholangitis and biliary obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Xi WU, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China